CLINICAL TRIAL: NCT03009058
Title: A Novel Phase I/IIa Open Label Study of IMM 101 in Combination With Selected Standard of Care (SOC) Regimens in Patients With Metastatic Cancer or Unresectable Cancer at Study Entry
Brief Title: Study of IMM 101 in Combination With Standard of Care in Patients With Metastatic or Unresectable Cancer
Acronym: MODULATE
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Commercial reasons
Sponsor: Immodulon Therapeutics Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IMM-101-011; 2016 001459 28 (EudraCT Number); CANC 32085 (Other: National Institute for Health Research (UK))
Record Dates: First submitted 2016-12-16; First posted 2017-01-04 (Estimated); Results first posted 2024-11-25 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-10

CONDITIONS: Metastatic Cancer
Keywords: Unresectable cancer; pancreatic; melanoma; breast; lung; colorectal; cholangio; sarcoma
MeSH Terms: conditions — Neoplasm Metastasis; Melanoma; Sarcoma | interventions — IMM-101; Gemcitabine; 130-nm albumin-bound paclitaxel; Albumin-Bound Paclitaxel; Capecitabine; Leucovorin; Fluorouracil; Irinotecan; Oxaliplatin; Cetuximab; spartalizumab; pembrolizumab; Nivolumab; Ipilimumab; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (17):
- IMM-101 + Gem panc ca (Experimental): IMM-101 will be given in combination with standard gemcitabine monotherapy. The treatment regimen with IMM-101 will be one dose given every 2 weeks for the first 3 doses followed by a rest period of 4 weeks, then one dose every 2 weeks for the next 3 doses. This is followed by a dose every 4 weeks thereafter.
  Interventions: Biological: IMM-101; Drug: Gemcitabine
- IMM-101+Gem/nab-paclitaxel panc ca (Experimental): IMM-101 will be given in combination with standard gemcitabine + nab-paclitaxel combination therapy.
  The treatment regimen with IMM-101 will be one dose given every 2 weeks for the first 3 doses followed by a rest period of 4 weeks, then one dose every 2 weeks for the next 3 doses. This is followed by a dose every 4 weeks thereafter.
  Interventions: Biological: IMM-101; Drug: Gemcitabine; Drug: Nab-paclitaxel
- IMM-101+Gem+capecitabine panc ca (Experimental): IMM-101 will be given in combination with gemcitabine + capecitabine combination therapy.
  The treatment regimen with IMM-101 will be one dose given every 2 weeks for the first 3 doses followed by a rest period of 4 weeks, then one dose every 2 weeks for the next 3 doses. This is followed by a dose every 4 weeks thereafter.
  Interventions: Biological: IMM-101; Drug: Gemcitabine; Drug: Capecitabine
- IMM-101 + FOLFIRINOX panc ca (Experimental): IMM-101 will be given in combination with standard FOLFIRINOX (FOLinic acid, Fluorouracil, IRINotecan and OXaliplatin) treatment.
  The treatment regimen with IMM 101 will be one dose given every 2 weeks for the first 3 doses followed by a rest period of 4 weeks, then one dose every 2 weeks for the next 3 doses. This is followed by a dose every 4 weeks thereafter.
  Interventions: Biological: IMM-101; Drug: Folinic Acid; Drug: Fluorouracil; Drug: Irinotecan; Drug: Oxaliplatin
- IMM-101+FOLFOX colorectal cancer (CRC) (Experimental): IMM-101 will be given in combination with standard FOLFOX (FOLinic acid, Fluorouracil and OXaliplatin) treatment.
  The treatment regimen with IMM-101 will be one dose given every 2 weeks for the first 3 doses followed by a rest period of 4 weeks, then one dose every 2 weeks for the next 3 doses. This is followed by a dose every 4 weeks thereafter.
  Interventions: Biological: IMM-101; Drug: Folinic Acid; Drug: Fluorouracil; Drug: Oxaliplatin
- IMM-101+FOLFIRI+CETUXIMAB colorectal cancer (CRC) (Experimental): IMM-101 will be given in combination with standard FOLFIRI (FOLinic acid, Fluorouracil and IRInotecan) + cetuximab combination treatment.
  The treatment regimen with IMM-101 will be one dose given every 2 weeks for the first 3 doses followed by a rest period of 4 weeks, then one dose every 2 weeks for the next 3 doses. This is followed by a dose every 4 weeks thereafter.
  Interventions: Biological: IMM-101; Drug: Folinic Acid; Drug: Fluorouracil; Drug: Irinotecan; Biological: cetuximab
- IMM-101+Gem cholangio (Experimental): IMM-101 will be given in combination with standard gemcitabine monotherapy. The treatment regimen with IMM-101 will be one dose given every 2 weeks for the first 3 doses followed by a rest period of 4 weeks, then one dose every 2 weeks for the next 3 doses. This is followed by a dose every 4 weeks thereafter.
  Interventions: Biological: IMM-101; Drug: Gemcitabine
- IMM-101+Gem lung ca (Experimental): IMM-101 will be given in combination with standard gemcitabine monotherapy. The treatment regimen with IMM-101 will be one dose given every 2 weeks for the first 3 doses followed by a rest period of 4 weeks, then one dose every 2 weeks for the next 3 doses. This is followed by a dose every 4 weeks thereafter
  Interventions: Biological: IMM-101; Drug: Gemcitabine
- IMM-101+Gem + nab-paclitaxel lung ca (Experimental): IMM-101 will be given in combination with standard gemcitabine + nab-paclitaxel combination therapy.
  The treatment regimen with IMM 101 will be one dose given every 2 weeks for the first 3 doses followed by a rest period of 4 weeks, then one dose every 2 weeks for the next 3 doses. This is followed by a dose every 4 weeks thereafter.
  Interventions: Biological: IMM-101; Drug: Gemcitabine; Drug: Nab-paclitaxel
- IMM-101+ anti-programmed death-1 (PD1) lung ca (Experimental): IMM-101 will be given in combination with standard treatment with either pembrolizumab or nivolumab.
  In order to ensure that there are no increased immune-related adverse events (AEs), the first 3 patients entering the anti-PD1 (pembrolizumab or nivolumab) cohort will receive IMM-101 at an increased dosing interval of every 4 weeks. In the absence of safety concerns for these patients after 3 doses of IMM-101, and following a robust safety review, all subsequent patients recruited to this treatment cohort will switch to the standard, more intensive (2-weekly induction dosing) IMM-101 dosing regimen.
  Interventions: Biological: IMM-101; Biological: Anti-PD1
- IMM-101+Gem melanoma (Experimental): IMM-101 will be given in combination with standard gemcitabine monotherapy. The treatment regimen with IMM-101 will be one dose given every 2 weeks for the first 3 doses followed by a rest period of 4 weeks, then one dose every 2 weeks for the next 3 doses. This is followed by a dose every 4 weeks thereafter.
  Interventions: Biological: IMM-101; Drug: Gemcitabine
- IMM-101+ anti-programmed death-1 (PD1) melanoma (Experimental): IMM-101 will be given in combination with standard treatment with either pembrolizumab or nivolumab. The first 3 patients entering the anti-PD1 (pembrolizumab or nivolumab) cohort will receive IMM-101 at an increased dosing interval of every 4 weeks. In the absence of safety concerns for these patients after 3 doses of IMM-101, and following a robust safety review, all subsequent patients recruited to this treatment cohort will switch to the standard, more intensive (2-weekly induction dosing) IMM-101 dosing regimen thereafter.
  Interventions: Biological: IMM-101; Biological: Anti-PD1
- IMM-101+ anti-cytotoxic T-lymphocyte associated protein 4 (CTLA-4) melanoma (Experimental): IMM-101 will be given in combination with standard treatment with ipilimumab. In order to ensure that there are no increased immune-related adverse events (AEs), the first 3 patients entering the ipilimumab cohort will receive IMM-101 at an increased dosing interval of every 4 weeks. In the absence of safety concerns for these patients after 3 doses of IMM-101, and following a robust safety review, all subsequent patients recruited to this treatment cohort will switch to the standard, more intensive (2-weekly induction dosing) IMM-101 dosing regimen thereafter.
  Interventions: Biological: IMM-101; Biological: Ipilimumab
- IMM-101+Gem breast cancer (Experimental): IMM-101 will be given in combination with standard gemcitabine monotherapy. The treatment regimen with IMM-101 will be one dose given every 2 weeks for the first 3 doses followed by a rest period of 4 weeks, then one dose every 2 weeks for the next 3 doses. This is followed by a dose every 4 weeks thereafter.
  Interventions: Biological: IMM-101; Drug: Gemcitabine
- IMM-101+Gem/ nab-paclitaxel breast (Experimental): IMM-101 will be given in combination with standard gemcitabine + nab-paclitaxel combination therapy.
  The treatment regimen with IMM-101 will be one dose given every 2 weeks for the first 3 doses followed by a rest period of 4 weeks, then one dose every 2 weeks for the next 3 doses. This is followed by a dose every 4 weeks thereafter.
  Interventions: Biological: IMM-101; Drug: Gemcitabine; Drug: Nab-paclitaxel
- IMM-101 + Gem sarcoma (Experimental): IMM-101 will be given in combination with standard gemcitabine monotherapy. The treatment regimen with IMM-101 will be one dose given every 2 weeks for the first 3 doses followed by a rest period of 4 weeks, then one dose every 2 weeks for the next 3 doses. This is followed by a dose every 4 weeks thereafter.
  Interventions: Biological: IMM-101; Drug: Gemcitabine
- IMM-101+cyclophosphamide (Experimental): IMM-101 will be given in combination with low dose cyclophosphamide (300mg/m2 in patients with solid malignancies.
  The treatment regimen with IMM-101 will be one dose given every 2 weeks for the first 3 doses followed by a rest period of 4 weeks, then one dose every 2 weeks for the next 3 doses. This is followed by a dose every 4 weeks thereafter.
  Interventions: Biological: IMM-101; Drug: Cyclophosphamide

INTERVENTIONS:
Biological: IMM-101 — A suspension of heat killed whole cell Mycobacterium obuense NCTC 13365
  Other Names: Heat killed M. obuense (NCTC 13365)
Drug: Gemcitabine — Standard of Care chemotherapy
  Other Names: GEMZAR
  Arms: IMM-101 + Gem panc ca; IMM-101 + Gem sarcoma; IMM-101+Gem + nab-paclitaxel lung ca; IMM-101+Gem breast cancer; IMM-101+Gem cholangio; IMM-101+Gem lung ca; IMM-101+Gem melanoma; IMM-101+Gem+capecitabine panc ca; IMM-101+Gem/ nab-paclitaxel breast; IMM-101+Gem/nab-paclitaxel panc ca
Drug: Nab-paclitaxel — Standard of Care chemotherapy
  Other Names: Abraxane
  Arms: IMM-101+Gem + nab-paclitaxel lung ca; IMM-101+Gem/ nab-paclitaxel breast; IMM-101+Gem/nab-paclitaxel panc ca
Drug: Capecitabine — Standard of Care chemotherapy
  Other Names: Xeloda
  Arms: IMM-101+Gem+capecitabine panc ca
Drug: Folinic Acid — Standard of Care chemotherapy
  Other Names: Leucovorin
  Arms: IMM-101 + FOLFIRINOX panc ca; IMM-101+FOLFIRI+CETUXIMAB colorectal cancer (CRC); IMM-101+FOLFOX colorectal cancer (CRC)
Drug: Fluorouracil — Standard of Care chemotherapy
  Other Names: 5FU
  Arms: IMM-101 + FOLFIRINOX panc ca; IMM-101+FOLFIRI+CETUXIMAB colorectal cancer (CRC); IMM-101+FOLFOX colorectal cancer (CRC)
Drug: Irinotecan — Standard of Care chemotherapy
  Other Names: Campto; Camptosar
  Arms: IMM-101 + FOLFIRINOX panc ca; IMM-101+FOLFIRI+CETUXIMAB colorectal cancer (CRC)
Drug: Oxaliplatin — Standard of Care chemotherapy
  Other Names: Eloxatin
  Arms: IMM-101 + FOLFIRINOX panc ca; IMM-101+FOLFOX colorectal cancer (CRC)
Biological: cetuximab — Standard of Care immunotherapy
  Other Names: Erbitux
  Arms: IMM-101+FOLFIRI+CETUXIMAB colorectal cancer (CRC)
Biological: Anti-PD1 — Standard of Care immunotherapy
  Other Names: pembrolizumab (KEYTRUDA),; nivolumab (OPDIVO)
  Arms: IMM-101+ anti-programmed death-1 (PD1) lung ca; IMM-101+ anti-programmed death-1 (PD1) melanoma
Biological: Ipilimumab — Standard of Care immunotherapy
  Other Names: YERVOY
  Arms: IMM-101+ anti-cytotoxic T-lymphocyte associated protein 4 (CTLA-4) melanoma
Drug: Cyclophosphamide — Standard of Care chemotherapy
  Other Names: cytophosphane
  Arms: IMM-101+cyclophosphamide

SUMMARY:
During this open label study patients will receive IMM-101 in conjunction with a recognised standard of care for metastatic or unresectable cancer for the patient's specific tumour type.

The primary objective of the study is to provide safety data for IMM-101 in combination with a number of selected standard of care regimens.

DETAILED DESCRIPTION:
The study will consist of three phases - Screening, Treatment and Maintenance. Patients who provide informed consent, will participate in a Screening period of up to 28 days to establish eligibility. Once eligibility is confirmed, patients will enter the Treatment Phase of the study.

In the Treatment Phase all patients will receive IMM-101 for 28 weeks.

At Week 32, if the Investigator considers it in the patients' best interest patients will progress to the Maintenance Phase of the study and will continue to be dosed every 4 weeks (or as close to this interval as permitted due to practical or logistical considerations). Patients will be followed up for assessment of safety, response to treatment, survival, and immunological markers for up to 4.5 years.

ELIGIBILITY:
Inclusion Criteria:

* Metastatic or unresectable cancer and considered by their physician to be indicated for a new line of SOC as listed in the protocol
* Are ineligible for a disease specific clinical study with IMM-101
* Have an estimated life expectancy greater than 3 months (from Day 0)
* Give signed informed consent for participation in the study
* Have an Eastern Cooperative Oncology Group (ECOG)/World Health Organisation (WHO) Performance Status of ≤2 at Day 0.
* Have adequate bone marrow, hepatic and renal function

Exclusion Criteria:

* Patient has previously received treatment with IMM-101
* Patient is currently part way through a course of chemotherapy or immunotherapy
* Patient is receiving concomitant treatment with another investigational product
* Patient has received an investigational drug within the 4 weeks prior to IMM 101 administration
* Patient has significant cardiovascular disease
* Patient has any previous or concurrent malignancy (excluding adequately treated carcinoma in situ of the cervix, basal cell carcinoma of the skin and/or non melanoma skin cancer, or if previous malignancy was more than 5 years prior to Screening and there are no signs of recurrence)
* Patient has co existing active infection or medical condition which will substantially increase the risk associated with the patient's participation in the study
* Patient has uncontrolled hypercalcaemia
* Patient has previously experienced an allergic reaction to any mycobacterial product.
* The patient has a history of non-infectious pneumonitis that required steroids or current pneumonitis
* Patient has received live vaccine within 30 days of planned start of study medication
* Patient is pregnant or a breast feeding woman.
* Patient is unwilling to use a medically acceptable, effective method of contraception throughout the treatment period and for at least 6 months after discontinuation of treatment.
* Patient has used depot corticosteroids in the 6 weeks before initiation of Screening
* Patient has had chronic use of systemic corticosteroids within the 2 week period before the first administration of IMM-101
* Patient has received a blood transfusion within 4 weeks prior to Screening
* In the opinion of the Investigator, the patient is unable or unwilling to comply with the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2017-05-31 (Actual); Primary Completion 2017-08-30 (Actual); Study Completion 2017-08-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Cunningham, MD FRCP, Principal Investigator — Royal Marsden Hospital Foundation Trust
Locations (4):
- France (2):
  - Centre Léon Bérard, Dpt Medecine & INSERM, Lyon
  - Gustave Roussy Cancer Center, Villejuif
- United Kingdom (2):
  - St George's University of London, Institute of Infection and Immunity, London
  - Royal Marsden Hospital Foundation Trust, London

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- IMM-101 in Combination With Anti PDL1 in Melanoma: Patients diagnosed with metastatic melanoma who were receiving an anti-programmed death (PD)-1 agent (nivolumab or pembrolizumab) therapy as standard of care were treated with IMM-101 in this cohort of the study.
Period: Overall Study
Arm/Group | IMM-101 in Combination With Anti PDL1 in Melanoma
Started | 2
Completed | 0
Not Completed | 2
Not completed — Study terminated soon after initiation for commercial reasons | 2

BASELINE CHARACTERISTICS:
Population: All enrolled patients
Groups:
- IMM-101 in Combination With Anti PDL1 in Melanoma: Patients diagnosed with metastatic melanoma who were receiving an anti-programmed death-1 (PD-1) agent (nivolumab or pembrolizumab) therapy as standard of care were treated with IMM-101 in this cohort of the study.
Arm/Group | IMM-101 in Combination With Anti PDL1 in Melanoma
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 1
Age, Continuous [Median (Full Range); unit: years] | 70 [63 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 2
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United Kingdom | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-related Adverse Events as Assessed by CTCAE v4.0
Description: Safety and tolerability will be measured by incidence and severity of adverse events (AEs), Laboratory abnormalities and local injection site reactions.
Time Frame: Due to the early termination of the study the outcome measure timeframe was until study termination, an average of 3 months.
Population: Both patients were assessed
Measure: Count of Participants; unit: Participants
Groups:
- IMM-101 in Combination With Anti PDL1 in Melanoma: Patients diagnosed with metastatic melanoma who were receiving an anti-PD-1 agent (nivolumab or pembrolizumab) therapy as standard of care were treated with IMM-101 in this cohort of the study.
Arm/Group | IMM-101 in Combination With Anti PDL1 in Melanoma
Number analyzed (Participants) | 2
Participants | 1

2. Secondary Outcome: Number of Participants With Treatment-related Adverse Events as Assessed by CTCAE v4.0
Description: Safety and tolerability will be measured by AEs, Laboratory abnormalities and local injection site reactions.
Time Frame: Week 28 through study completion (maximum 4.5 years)
Population: Study was terminated before the Week 28 timepoint was reached.
Groups:
- IMM-101 in Combination With Anti PDL1 in Melanoma: Patients diagnosed with metastatic melanoma who were receiving an anti-PD-1 agent (nivolumab or pembrolizumab) therapy as standard of care were treated with IMM-101 in this cohort of the study.
  A minimum of 10 patients per cohort were required for an evaluation of futility with respect to the primary activity endpoint of response to treatment (based on immune-related response criteria [irRC]). Given that only two patients were enrolled into the study, the objectives of the study described in the study protocol cannot be met.
Arm/Group | IMM-101 in Combination With Anti PDL1 in Melanoma
Number analyzed (Participants) | 0

3. Secondary Outcome: Number of Participants With Treatment-related Adverse Events When IMM-101 is Given in Combination With a Checkpoint Blockade Inhibitor
Description: Safety and tolerability will be measured by AEs, Laboratory abnormalities and local injection site reactions to evaluate whether there is any exacerbation of toxicity normally observed with these agents
Time Frame: From screening until study termination an average of 3 months.
Population: Both patients enrolled
Measure: Count of Participants; unit: Participants
Arm/Group | IMM-101 in Combination With Anti PDL1 in Melanoma
Number analyzed (Participants) | 2
Participants | 1

4. Secondary Outcome: Response to Treatment
Description: Response to treatment, (defined as immune related Stable Disease (irSD), immune related Partial Response (irPR) and immune related Complete Response (irCR) as assessed by the Investigator:
  * Immune-related Complete Response (irCR) is the disappearance of all lesions, measured or unmeasured, and no new lesions
  * Immune-related Partial Response (irPR) is a ≥50% drop in tumour burden from baseline as defined by the irRC
  * Immune-related Progressive Disease (irPD) is ≥25% increase in tumour burden from the lowest level recorded.
  * Everything else is considered immune-related Stable Disease (irSD).
Time Frame: Per protocol the initial assessment was at Week 28 then through study completion (maximum 4.5 years). Due to early termination of the study, response to treatment was measured at Week 11 for both patients
Measure: Count of Participants; unit: Participants
Arm/Group | IMM-101 in Combination With Anti PDL1 in Melanoma
Number analyzed (Participants) | 2
Participants
  immune related Stable Disease [irSD] | 1
  immune related Partial Response [irPR] | 1
  immune related Complete Response [irCR] | 0

5. Secondary Outcome: Overall Survival (OS)
Description: Assessment of overall survival (defined as the time from enrolment to death due to any cause).
Time Frame: From date of randomization until date of first documented progression or date of death from any cause, whichever came first, assessed up to 60 months.
Population: Assessment of overall survival (defined as the time from enrolment to death due to any cause). However, whilst 2 participants were monitored and analyzed, neither patient died before the study was terminated.
Measure: Count of Participants; unit: Participants
Arm/Group | IMM-101 in Combination With Anti PDL1 in Melanoma
Number analyzed (Participants) | 2
Participants | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time of consent until 28(±7 days) received at week 10 date which is around 3 months after the last dose of IMM-101. Serious Adverse Events were followed to resolution irrespective of the date of the last dose
Description: Adverse events (including those reported spontaneously by the patient or observed by the Investigator) were recorded from the time of informed consent. All adverse events were followed until resolution, death or 30 days after the End of Study/Withdrawal visit (whichever came first). Study treatment related serious adverse events (SAEs) were recorded regardless of time from last dose.
Arm/Group | IMM-101 in Combination With Anti PDL1 in Melanoma
All-Cause Mortality (participants affected / at risk) | 0/2
Serious Adverse Events (participants affected / at risk) | 0/2
Other Adverse Events (participants affected / at risk) | 1/2
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IMM-101 in Combination With Anti PDL1 in Melanoma (N=2)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) — Head pain (at site of biopsy)
Hyperthyroidism (Endocrine disorders) | 1 (1) — Subclinical hyperthyroid
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Only two patients were enrolled into the study before the study was terminated early by the Sponsor for commercial reasons. There were no specific safety concerns based on the data from the two patients treated. These limited data provide some preliminary indication regarding the safety and tolerability of IMM-101 when administered in combination with nivolumab. No meaningful assessment of efficacy could be made given that only two patients were enrolled into the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2016-10-25): https://cdn.clinicaltrials.gov/large-docs/58/NCT03009058/Prot_000.pdf
  • Statistical Analysis Plan (2017-09-26): https://cdn.clinicaltrials.gov/large-docs/58/NCT03009058/SAP_001.pdf